CLINICAL TRIAL: NCT04705883
Title: Vaginal Prasterone In The Treatment Of Vaginal Atrophy In Patients With Breast Cancer Treatment With Aromatase Inhibitors (Vibra Study)
Brief Title: Vaginal Prasterone In Vaginal Atrophy In Breast Cancer Survivors
Acronym: VIBRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Camil Castelo-Branco, Principal Investigator, Clinical Professor, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Versión 4- 20/09/2020
Record Dates: First submitted 2021-01-11; First posted 2021-01-12 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Vulvar Atrophy; Breast Cancer; Genitourinary Syndrome of Menopause
Keywords: Breast Cancer; Genitourinary Syndrome of Menopause
MeSH Terms: conditions — Breast Neoplasms | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prasterone (Other): 10 patients will be treated using prasterone during 6 months.
  Interventions: Drug: Prasterone (DHEA), Micronized

INTERVENTIONS:
Drug: Prasterone (DHEA), Micronized — Vaginal prasterone 6,5mg/24h first month, next 5 months 6,5mg/48h, vaginal administration.
  Other Names: Intrarosa

SUMMARY:
VAGINAL PRASTERONE in the treatment of VAGINAL ATROPHY IN PATIENTS WITH BREAST CANCER TREATMENT WITH AROMATASE INHIBITORS (VIBRA STUDY)

DETAILED DESCRIPTION:
Verify a clinical improvement of AVV without increasing levels of ultrasensitive blood estradiol in breast cancer survivors treated with aromatase inhibitors by administering vaginal prasterone.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer treated with anti-hormonal therapy based on inhibitors of aromatase (IA) (letrozole, anastrozole or exemestane) ± analogues of the GnRH (aGnRH)
* Menopause (natural or induced) and signs / symptoms of vulvovaginal atrophy
* Cytology and / or determination of Human Papillomavirus (HPV) negative
* Intention or willingness to have sex

Exclusion Criteria:

* To have received topical hormonal treatment in the last 6 months or Have used vaginal moisturizers and / or lubricants during the 30 days prior to the study treatment
* To have received treatment with laser, radiofrequency, hyaluronic acid, etc. in the vagina during the last two years at the beginning of the study
* To Have: an active infection of the genital tract; an intraepithelial neoplasm of the cervix, vagina or vulva; suspected of suffering or having been treated for cancer of the genital tract; suffer a genital prolapse of II degree or greater

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Estradiol | 12 months
  Ultrasensitive blood estradiol, serum levels measured in pg/ml

SECONDARY OUTCOMES:
Vaginal pH | 12 months
  vaginal pH measured by ph roll from 1 to 14 (the lesser the better)
Vaginal maturation index | 12 months
  vaginal maturation index meadured by vaginal citology on percentage from 0 to 100 divided in superficial, intermediate and basal cells. The more superficial, the better.
Vaginal health index | 12 months
  To describe if there is a correlation between changes in the visual examination of the vagina. using the vaginal health index: from 5 to 25 (min-max). The higher the better.
Female Sexual Function Index | 12 months
  Questionaire from 18 to 90 (min-max). The higher the better.
Social Functioning Questionnaire | 12 months
  Questionaire Social Functioning 12 (Physical and Mental Health Composite Scores) from 0 to 12 (min-max). The higher the better.

CONTACTS AND LOCATIONS:
Overall Officials: Camil Castelo-Branco, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No